CLINICAL TRIAL: NCT05392166
Title: Prevalence and Factors Associated With Pancreatic Enzyme Elevations Among Children With Type 1 Diabetes Hospitalized With Diabetic Ketoacidosis
Brief Title: Prevalence and Factors Associated With Pancreatic Enzyme Elevations Among Diabetic Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Walaa Saber Kassem, resident doctor at pediatric department at faculty of medicine sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-22-05-09
Record Dates: First submitted 2022-05-15; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Children
MeSH Terms: interventions — Blood Gas Analysis; Blood Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case (Active Comparator)
  Interventions: Diagnostic Test: blood glucose, blood gases, serum electrolytes, HbA1c, complete blood count and serum creatinine. Serum calcium, serum amylase, serum lipase and serum triglycerides , abdominal ultrasound
- control (Active Comparator)
  Interventions: Diagnostic Test: blood glucose, blood gases, serum electrolytes, HbA1c, complete blood count and serum creatinine. Serum calcium, serum amylase, serum lipase and serum triglycerides , abdominal ultrasound

INTERVENTIONS:
Diagnostic Test: blood glucose, blood gases, serum electrolytes, HbA1c, complete blood count and serum creatinine. Serum calcium, serum amylase, serum lipase and serum triglycerides , abdominal ultrasound — blood samples will be collected at admission for assessment of blood glucose, blood gases, serum electrolytes, HbA1c, complete blood count and serum creatinine. Serum calcium, serum amylase, serum lipase and serum triglycerides will be assessed within the first 24 hours after hospital admission. For the control group, the blood samples will be collected during the pediatric diabetes clinic follow-up visits. Abdominal ultrasound will be done to all the study participants.

SUMMARY:
Acute pancreatitis was reported as a DKA associated complication. The true incidence and clinical significance of pancreatitis in children with DKA is unclear. And its diagnosis in children requires a high index of clinical suspicion . Severe hypertriglyceridemia is an uncommon T1D complication which is also due to insulin deficiency and which can trigger acute pancreatitis The triad of DKA, severe hypertriglyceridemia, and acute pancreatitis have been described in children, especially in those with new onset T1D, abdominal pain and vomiting occasionally prompt the measurement of pancreatic enzymes Previous studies indicate that pancreatic enzyme elevations, particularly increased serum lipase levels, are very common in children with DKA. The magnitude of lipase elevation appears to correlate with the degree of acidosis, whereas increased serum amylase level is nonspecific. The majority of patients with elevated enzymes had no significant abdominal symptoms or delay in their clinical recovery. In those with persistent abdominal symptoms after acidosis resolved, abdominal CT findings were normal. The results of previous pediatric studies were comparable to those from studies in adult patients with DKA. Amylase and/or lipase elevations have been reported in 24.7% to 79% of cases. However, the incidence of acute pancreatitis in DKA seems to be higher in adults compared with children and is reported to be more than 10% they also have found that pancreatic enzyme elevations occur much less commonly in the setting of new-onset diabetes without DKA. Consistent with this observation, pancreatic enzymes have been reported to be higher in patients with poorly controlled diabetes compared with those in good control. It was postulated to result from direct injury to the pancreas with enzyme leakage from the acini, secretion of amylase and lipase from non-pancreatic sources, and decreased renal clearance .Acute pancreatitis also is attributed to hypertriglyceridemia.

the diagnosis of Acute Pancreatitis requires 2 of the 3 criteria: (1) abdominal pain not due to other causes, (2) elevated serum lipase or amylase 3 times the upper limit of the normal reference range (ULN), and/or (3) imaging evidence of pancreatitis . But also, there are limitations associated with each criterion in children . Although abdominal pain is the most common presentation, up to one third of patients may not report abdominal pain and radiation of pain to the back occurs in5% .

ELIGIBILITY:
Inclusion Criteria:

- children aged 0-12 years, diagnosed with type 1 diabetes mellitus and admitted to the pediatric emergency department with DKA criteria including, Blood glucose level > 200 mg/dl, pH < 7.3, and /or bicarbonate level in blood < 15 mmol/l and positive ketones in urine by dipstick method, will be included. Age, sex and duration of diabetes matched control children without DKA will be recruited from T1DM children attending the pediatric diabetes clinic at Sohag university hospital.

Exclusion Criteria:

* Patients diagnosed with congenital or acquired chronic pancreatitis or gall stones will be excluded.

Ages: 1 Day to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-05-13 (Estimated); Study Completion 2023-05-13 (Estimated)

PRIMARY OUTCOMES:
pancreatic enzymes elevation in diabetic children . | 1year
  assesment of level of serum amylase and serum lipase within 24 hours of admission

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sharma PK, Kumar M, Yadav DK. Severe Hypertriglyceridemia Causing Pancreatitis in a Child with New-onset Type-I Diabetes Mellitus Presenting with Diabetic Ketoacidosis. Indian J Crit Care Med. 2017 Mar;21(3):176-178. doi: 10.4103/ijccm.IJCCM_281_16. PMID 28400692
- [Background] Wolfgram PM, Macdonald MJ. Severe Hypertriglyceridemia Causing Acute Pancreatitis in a Child with New Onset Type I Diabetes Mellitus Presenting in Ketoacidosis. J Pediatr Intensive Care. 2013;2(2):77-80. doi: 10.3233/PIC-13053. PMID 24455446
- [Background] Saengkaew T, Sahakitrungruang T, Wacharasindhu S, Supornsilchai V. DKA with Severe Hypertriglyceridemia and Cerebral Edema in an Adolescent Boy: A Case Study and Review of the Literature. Case Rep Endocrinol. 2016;2016:7515721. doi: 10.1155/2016/7515721. Epub 2016 Jan 20. PMID 26904318
- [Background] Radhakutty A, Shen J, Hooper AJ, Miller SA, Burnett JR, Mah PM, Burt MG, Doogue MP. Quantification and genotyping of lipoprotein lipase in patients with diabetic lipaemia. Diabet Med. 2014 Dec;31(12):1702-7. doi: 10.1111/dme.12565. Epub 2014 Sep 17. PMID 25131724